CLINICAL TRIAL: NCT00245401
Title: CYPHERTM Stent Post-Marketing Surveillance Registry (US-PMS)
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Cordis US Corp. (Industry)
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: P03-6321
Record Dates: First submitted 2005-10-04; First posted 2005-10-28 (Estimated); Last update posted 2007-04-04 (Estimated); Status verified 2007-04

CONDITIONS: Coronary Artery Disease
MeSH Terms: conditions — Coronary Artery Disease

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

INTERVENTIONS:
Device: CYPHERTM Sirolimus-Eluting Coronary Stent

SUMMARY:
The purpose of this PMS registry, named e-CYPHER Stent Registry, is to collect post marketing surveillance data on the CYPHERTM Sirolimus-eluting Coronary Stent following marketing approval, when used in normal clinical practice within the labeled indications.

ELIGIBILITY:
Inclusion Criteria:

* Cypher stent

Exclusion Criteria:

* N/A

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 2070
Dates: Start 2003-08; Study Completion 2004-12 (Actual)

PRIMARY OUTCOMES:
MACE at 30 days, 6 months and 1 year.

SECONDARY OUTCOMES:
There is no pre-specified secondary outcome.

CONTACTS AND LOCATIONS:
Overall Officials: Emerson Perin, MD, Principal Investigator — Texas Heart Institute

REFERENCES:
- [Derived] Bezerra H, Perin E, Berger P, Block P, Ramee S, Katz S, Kellet M, Dippel E, Schaer G, Britto S, Cohen S, Costa M. Outcomes of unselected recipients of sirolimus-eluting stents: the Cypher stent U.S. post-marketing surveillance registry. J Invasive Cardiol. 2010 Feb;22(2):48-55. PMID 20124586